CLINICAL TRIAL: NCT04109326
Title: Effect of a Tailored Program of Physical Activity and Nutritional Therapeutic Education on Clinical, Psychological and Sociological Factors in Breast Cancer Patients Undergoing Adjuvant Treatment : Multicenter Randomized Controlled Trial
Brief Title: Effect of a Program of Physical Activity and Nutritional Therapeutic Education in Breast Cancer Patients
Acronym: APAD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VA2012/39; 2012-A01648-35 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Physical activity; Nutrition; Therapeutic education; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — 3-acetylpyridine adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: * The experimental arm "APAD": tailored PA program associated with individual nutritional counseling whilst hospitalization and at home during the 26-week duration of adjuvant treatment
  * The control arm: standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity and Dietetique (Experimental): tailored PA program associated with individual nutritional counseling whilst hospitalization and at home during the 26-week duration of adjuvant treatment
  Interventions: Other: APAD
- Control (No Intervention): Standard of care

INTERVENTIONS:
Other: APAD — 8 PA sessions supervised at the hospital centers and 44 unsupervised home sessions, to be performed twice a week.
  6 consultations for nutrition education to teach the principles of well balanced diet, to foster weigh control during treatment, and to induce appropriate feeding behaviors after treatment.
  Arms: Adapted Physical Activity and Dietetique

SUMMARY:
This multicenter randomized controlled trial aims to evaluate the effect of a tailored program of physical activity and nutritional therapeutic education on clinical, psychological and sociological factors in breast cancer patients undergoing adjuvant treatment.

DETAILED DESCRIPTION:
The experimental arm "APAD": tailored PA program associated with individual nutritional counseling whilst hospitalization and at home during the 26-week duration of adjuvant treatment

The experimental program will include:

* 8 PA sessions supervised at the hospital centers and 44 unsupervised home sessions, to be performed twice a week.
* 6 consultations for nutrition education to teach the principles of well balanced diet, to foster weigh control during treatment, and to induce appropriate feeding behaviors after treatment.

The control arm: standard of care

ELIGIBILITY:
Inclusion Criteria:

* Female patient with histologically proven breast cancer
* Age ≥18 years old
* Patients having undergone curative surgery and eligible to 6 cycles of adjuvant chemotherapy (6 FEC100, or 3FEC100 + 3 taxanes) followed by radiotherapy
* Satisfactory healing from surgical act on breast and lymph nodes
* Ability to understand the nature, goal and study methodology
* Consent to cooperate for clinical assessments
* Affiliation to a social security regime or beneficiary of equivalent social protection
* Written informed consent provided before any study specific procedures

Exclusion Criteria:

* Metastatic disease
* Any other primary tumor
* Contra-indication to moderate physical activity: Unchecked high blood pressure; family history of sudden death in a first degree relative; not stabilized heart disease; acute or chronic lung disease resulting in dyspnea for moderate effort; uncontrolled diabetes, carrying a stent; other severe pathologies unstabilized, disabled or not indicated to physical practice.
* Contra-indication to adjuvant chemotherapy or radiotherapy
* Pregnancy or breast feeding (according to the recommendations of the usual adjuvant breast cancer)
* Inability to attend or comply with interventions or follow-up scheduling, disability or difficulty preventing a proper understanding of trial instructions
* Legal inability or restricted legal ability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2016-01-05 (Actual); Study Completion 2016-06-11 (Actual)

PRIMARY OUTCOMES:
Rate of cancer-related fatigue | 6 months
  The primary assessment criterion is subjective fatigue measured using the 'General Fatigue' subscale of the Multidimensional Fatigue Inventory (MFI-20) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Romieu, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (8):
- France (8):
  - Institut Sainte Catherine, Avignon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CH Ambroise Paré, Marseille
  - CH Montélimar, Montélimar
  - ICM, Montpellier
  - Centre Eugène Marquis, Rennes
  - Institut de Cancéologie de l'Ouest, Saint-Herblain